CLINICAL TRIAL: NCT03644355
Title: Obesity and Asthma: Determinants of Inflammation and Effect of Intervention
Brief Title: Asthma and Obesity Diet Versus Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Melinda Sothern, Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSUHSC IRB 7437
Record Dates: First submitted 2018-06-25; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity, Childhood; Asthma in Children; Inflammatory Response; Metabolic Syndrome; Nutrition Poor; Physical Activity; Behavior, Eating; Molecular Biology, Restriction Fragment Length Polymorphisms; Maternal Exposure; Genetic Change
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome; Malnutrition; Motor Activity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Cross-sectional, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diet and Nutrition Education (Experimental): Lifestyle counseling plus nutrition education and counseling and protein sparing modified fast diet plus supplementation of vitamins and minerals, followed by a balanced, hypo-caloric diet and nutrition education provided by a registered dietician
  Interventions: Behavioral: Lifestyle counseling
- Exercise Instruction (Active Comparator): Lifestyle counseling plus moderate intensity, progressive exercise prescription including cardio-pulmonary, strength and flexibility exercise tailored to the individual needs of each participant.
  Interventions: Behavioral: Lifestyle counseling
- Combined Diet and Exercise (Active Comparator): Lifestyle counseling plus dietary intervention including nutrition education and counseling and a protein sparing modified fast diet and nutrition education combined with the exercise intervention including a moderate intensity, progressive exercise prescription including cardio-pulmonary, strength and flexibility exercise tailored to the individual needs of each participant.
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention): Delayed intervention (waiting list) group receives no intervention for 12 weeks followed by the Diet plus Exercise intervention.

INTERVENTIONS:
Behavioral: Lifestyle counseling — Inter-disciplinary, interactive, family based behavioral intervention for overweight children
  Other Names: Trim Kids Behavioral Counseling Intervention
  Arms: Combined Diet and Exercise; Diet and Nutrition Education; Exercise Instruction

SUMMARY:
Obesity is recognized as a pro-inflammatory condition associated with multiple chronic diseases, including asthma. The specific mechanisms linking asthma and obesity remain hypothetical. Our primary hypothesis is that inflammatory SNPs may regulate the degree of the inflammatory response, with obesity modifying the severity of the disease. In this instance, asthma that develops in the context of obesity demonstrates the potential deleterious relationship between a specific proinflammatory state (obesity) and the genetic regulators of inflammation (SNPs). Our secondary hypothesis proposes that short-term (12-weeks) weight loss by diet alone, but not exercise alone, will reduce lung specific inflammation and diminish the pro-inflammatory responses in female African American obese adolescents with asthma compared to a waiting list control group who after their initial 12 weeks then receive a combined 12-week diet plus exercise program (waiting list control/combined). A third exploratory hypothesis proposes that the frequency of identified SNPs will be significantly related to the amount of fat loss through diet, exercise or combined program and will further be mediated by specific airway and, pro-and-anti-inflammatory markers.These hypotheses will be tested using the following Specific Aims:

1. To determine the frequency of single nucleotide polymorphisms and SNP haplotypes in pro- and anti-inflammatory genes in female African American obese and non-obese asthmatic and non-asthmatic adolescents, 13-19 years or age.
2. To examine the effects of diet or exercise on lung specific inflammation (exhaled nitric oxide, [eNO]) and pro-and-anti-inflammatory responses in female African-American obese asthmatic and non-asthmatic adolescents compared to a waiting list control/ combined group.

In addition we will examine the following Exploratory Aim:

To determine the effects of the inflammatory SNPs in the modulation of several inflammatory markers and lung specific inflammation (eNO) in female African-American obese asthmatic and non-asthmatic adolescents before and after weight loss through diet, exercise or both.

DETAILED DESCRIPTION:
Our primary hypothesis is that inflammatory SNPs may regulate the degree of the inflammatory response, with obesity modifying the severity of the disease. In this instance, asthma that develops in the context of obesity demonstrates the potential deleterious relationship between a specific proinflammatory state (obesity) and the genetic regulators of inflammation (SNPs).

Our secondary hypothesis proposes that short-term (12-weeks) weight loss by diet alone, but not exercise alone, will reduce lung specific inflammation and diminish the pro-inflammatory responses in female African American obese adolescents with asthma compared to a waiting list control group who after their initial 12 weeks then receive a combined 12-week diet plus exercise program (waiting list control/combined). A third exploratory hypothesis proposes that the frequency of identified SNPs will be significantly related to the amount of fat loss through diet, exercise or combined program and will further be mediated by specific airway and, pro-and-anti-inflammatory markers. Specific aims include:

1. To determine the frequency of single nucleotide polymorphisms and SNP haplotypes in pro- and anti-inflammatory genes in female African American obese and non-obese asthmatic and non-asthmatic adolescents, 13-19 years or age.
2. To examine the effects of diet or exercise on lung specific inflammation (exhaled nitric oxide, [eNO]) and pro-and-anti-inflammatory responses in female African-American obese asthmatic and non-asthmatic adolescents compared to a waiting list control/ combined group.
3. To determine the effects of the inflammatory SNPs in the modulation of several inflammatory markers and lung specific inflammation (eNO) in female African-American obese asthmatic and non-asthmatic adolescents before and after weight loss through diet, exercise or both.

We will conduct a cross-sectional analysis of 4 groups of African American adolescent (13-19 years) females as follows: Group 1A: Obese with asthma Group 1B: Non-obese with asthma Group 1C: Obese non-asthmatics Group 1D: Non-obese, non-asthmatics

Patients included in this part of the study will be female African American obese and non-obese asthmatic adolescents, 13-19 years, as defined by United States Centers for Disease control (USCDC 2000 sex specific Body Mass Index (BMI)-for-age growth charts. As controls we will include female African American obese, non asthmatic adolescents and healthy age matched controls (non-obese, non-asthmatics).

Assuming a dominant model, for a haplotype of 5 SNPs, a sample of 100 individuals per group (matching 1:1) would achieve at least 80% power to detect an OR of 1.5 for the association of the haplotype with group membership (such as obese with asthma vs. non-obese with asthma), at 0.05 significance level. All other group comparisons would assume the same conditions, thus samples of 100 for each of the groups are required.

After parent/guardian has signed the informed consent, a general medical exam and history is taken, and spirometry testing is performed to assess the lung function of each participant, obesity status will be assessed. For girls found to be non-obese during visit 1, approximately 30 ml of peripheral blood will be obtained from 100 asthmatics and 100 non-asthmatic healthy age matched controls. For obese participants (100 asthmatic and 100 non-asthmatics), peripheral blood draws will be obtained during visit 2 (baseline). Peripheral blood will be tested for a Hemoglobin A1-C (HA1C), lipid profile and to determine the presence of inflammation and genetic markers. An additional blood sample from all African American adolescent girls participating in the study will be collected into heparin tubes (2 10ml tubes). The mononuclear layer will be separated using density gradients and will characterize the circulating MDS. Flow cytometry will be used to determine the percentage of monocytic or granulocytic MDSC using several fluorescence-labeled antibodies, including anti-CD11b, CD14, CD15, CD33, CD66 and HLA-DR. The DNA will be extracted by DNAzol (Invitrogen Corp; Grand Island, NY). For the SNP analysis we plan to use the humanCNV370-Quad bead chip from lllumina (lllumina Inc, San Diego, CA). This chip allows the analysis of more than 370,000 SNPs simultaneously and uses only 200 ng of genomic DNA. We will initially focus our analysis in the pro- and anti-inflammatory cytokine gene SNPs (/LS, TNF, TGFB, ILIO, IL8, IL6, PTGS2, ARG1) and SNPs in leptin, leptin receptor and adiponectin (Table 11) and the results will be confirmed by TaqMan as follows: genomic DNA (5 ng) will be denatured at 95°C for 10 min and amplified for 40 cycles of 15 sec at 92°C and 1 min at 58°C, in the presence of 2X TaqMan Universal Master Mix (Applied Biosystems), water, and the respective primer and reporter probe mix (labeled with either FAM or VIC). The reaction will be analyzed using a 7900 HT instrument (Applied Biosystems), for the presence of VIC or FAM fluorescence marker, or both, using the Sequence Detection System (Applied Biosystems) to determine the genotype. Controls will include individuals of known genotype and blanks without DNA. In addition, 15% of the samples will be run twice in separate assays and the allele classification compared. The individuals of known genotype and blanks without DNA will be included for each SNP in every batch.

Chi-square, Fisher's exact, and student-t tests will be used to assess the statistical significance of the differences in the frequencies of the different SNPs between obese asthmatics, non-obese asthmatics, obese non-asthmatics and healthy controls. Haplotype frequencies will be inferred using log-linear modeling embedded within an expectation-maximization algorithm. Quality control procedures (including evaluation of genotyping efficiency and Hardy-Weinberg equilibrium), assessment of linkage disequilibrium between markers as well as haplotype association analysis will be performed separately in obese versus nonobese and asthmatic versus non-asthmatics.

After enrollment, eligible participants will undergo a baseline visit to include approximately 30ml peripheral blood draw, Dual Energy X-RAY Absorptiometry (DEXA) scan, exhaled nitric oxide (eNO), and study eligibility per the study physician. Following this baseline visit, obese participants with and without asthma will be randomized to:

1) diet only, 2) exercise only or 3) waiting list/combined intervention (no intervention for 12 weeks followed by combined diet and exercise).

Approximately 110 subjects will be recruited per treatment and control group. Assuming an attrition rate of 20%, we will maintain 360 subjects, 90 per group which will provide adequate statistical power to:

1. detect significant differences in eNO between diet only, exercise only, combined program, or a waiting list control group of female African American obese asthmatics and non-asthmatics as per the sample size power calculations below and;
2. as part of the exploratory aim 3, determine the effects of the inflammatory SNPs in the modulation of inflammatory markers and eNO in female African-American obese asthmatic and non-asthmatic adolescents before and after weight loss through diet, exercise or both as per the sample size power calculations).

Intervention Methods:

Treatment groups will receive the Trim Kids behavior modification program but the intervention materials will be specific to diet only or exercise only treatments. Non-obese asthmatics and non-obese, non-asthmatics will serve as controls for the exploratory aim and participate in a general medical exam, spirometry and blood testing only. Parents and children attend a weekly two-hour comprehensive session for a recommended time period. Medical supervision and guidance are provided by a physician or nurse at each session in order to increase compliance and monitor side effects.

Management of asthma: We will exclude persons with severe or uncontrolled asthma. In the case of acute asthma attacks participants will be managed according to a written and reviewed asthma action plan, with the use of asthma medications or S-agonists like Albuterol, and if necessary with a short course of other medications. Asthmatic participants involved in the intervention group will also be required to use a pre-exercise dose of asthma medication before participation in each exercise session or will be excluded from that session. Any exacerbation will be recorded and participants will be able to contact a health provider, and if needed will be referred to emergency services. In case of a more severe exacerbation or progressive worsening, the participant will be treated according to standard of care, and taken off the study if chronic or prolonged anti-inflammatory treatment is considered a priority.

Nutrition education includes a series of learning activities, which are specific to needs of each group as they progress through the different stages of the treatment program. The children are provided with easy-to-use food frequency checklists to fill in each week.

The exercise protocols to be utilized in this study will be based on the Trim Kids exercise protocol, which tailors the recommendations to the child's medical condition (co-morbidities such as asthma), weight status and fitness level. All exercise recommendations will follow the guidelines of the American Thoracic Society (ATS), American Academy of Pediatrics (AAP) and American Academy of Sports Medicine (ACSM). Exercise sessions at the LSUHSC Wellness center will be supervised by ACSM certified instructors and personal trainers. During each 12-week session of the program, the exercise activities correspond with the group's physical condition of obesity and ability to comprehend, synthesize and apply health and fitness Information to daily life situations. Children receive an exercise video containing an exercise routine to perform at home. They are also given cards to record the number of minutes of physical activity, they perform each week. Compliance is monitored by observing these physical activity record cards and monitoring of heart and breathing rate. Behavior modification and psychosocial education are integrated into educational sessions by a psychologist.

Behavior modification skills are taught stressing how discussion, modeling, role playing and guided problem solving are used. Topics such as self-monitoring, commitment, limit setting, habit formation, goal setting and action plans, decision-making skills and assertiveness training are discussed.

The intervention will be conducted at the Louisiana State University (LSU) Health Sciences Center Wellness Facility. Both diet and exercise groups will meet for medical monitoring and weigh in a clinical area adjacent to a private room with a scale during the first 30 minutes of each weekly class.

The diet only group will meet in a classroom after the 30-minute medical monitoring and weigh-in. Behavior modification class will follow for 30 minutes and Nutrition education for approximately 30-60 minutes. Study participants enrolled in the diet only intervention will be placed on either a protein modified fast diet plus supplementation of vitamins and minerals, followed by a balanced, hypo-caloric diet and/or a moderate intensity, progressive exercise program, and given instruction on behavior modification.

The exercise only group will meet in the large multi-purpose room after the 30 minute medical monitoring and weigh in. Behavior modification class will follow for 30 minutes. Participants will utilize the aerobic equipment, attend culturally specific dance classes, participate in strength training, and outdoor family field sports in an adjacent community park area for approximately 30-60 minutes. The participants exercise in a playful, sporadic, intermittent manner while the instructor discusses key concepts using symbols, music and various props.

Following a 12 week waiting period, participants in the combined program will meet in a separate multi-purpose room and will participate in diet, exercise and behavior modification sessions once per week.

ELIGIBILITY:
Inclusion Criteria:

* African American Females with an age of 13-19 years will be recruited. Our aim is to target high school age youth who are most likely to exhibit autonomy and authority to control both their nutrition and exercise regimens. In addition this age range is representative of the age group most likely to access school based health centers for recruitment purposes. Lastly, the study includes the collection of blood samples for the purpose of examining varied physiologic parameters that are affected by maturation. Participants above the age of 13 are most likely pubertal and thus, less likely to be affected by maturation issues.

Exclusion Criteria:

* Presence of other chronic pulmonary or systemic disease.
* Presence of moderate or severe atopic dermatitis or allergic rhinitis.
* Severe asthmatic based upon American Thoracic Society (ATS) standards and/or NIH guidelines.
* Acute lower respiratory infection in the last 2 weeks before baseline eNO evaluation.
* Pregnant are nursing mothers Study participants and parents (s) will be advised of the known risks and consequences associated with the testing and also of the reasonably known risks and consequences of not undergoing testing.

Severe or uncontrolled asthmatics will not be allowed to participate.

Participants with a recent (in the last 2 weeks) lower respiratory infection will not be allowed to participate.

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

PRIMARY OUTCOMES:
exhaled nitric oxide, [eNO] change | Baseline visit and and post intervention at 13 to 15 weeks
  Exhaled nitric-oxide (eNO; to be performed at baseline visit and post intervention at 13 to 15 weeks):
  The eNO level will be measured by chemiluminescence gas analyzer (Niox®), standardized according to the American Thoracic Society guidelines, 1999 [29]. NO is produced in healthy airway for normal physiologic functions (maintaining airway patency). It is formed during airway inflammation and may contribute to oxidative stress. It is overproduced in the lungs of asthmatic patient. Evidence suggests that eNO may be used as marker for lung inflammation [30-33; 112].

SECONDARY OUTCOMES:
Body Mass Index Change | Baseline visit and and post intervention at 13 to 15 weeks
  Body Mass Index (BMI) will be calculated from weight and height measurements at the baseline visit and post intervention at 13 to 15 weeks. The BMI is the weight in kilograms divided by the square of the height in meters. BMI will be evaluated using the 2000 CDC-BMI for age growth charts [102]. Consensus classifies those children with BMI >95*^ percentile as obese.
Single nucleotide polymorphisms (SNPs) | Baseline clinical visit
  Analyzed from a blood sample, using the lllumina system
Arginase activity | Baseline clinical visit
  Arginase activity will be determined as described before. Briefly, twenty five microliters of serum will be mixed with 25 µl of 50 mM Tris-HCl, pH 7.5, containing 10 mM MnCl2, and incubated at 55°C for 10 min to activate the enzyme. One hundred fifty microliters of 100 mM carbonate buffer and 50 µl of 100 mM L-arg will be added and the samples incubated at 37°C for 20 min. The reaction will be stopped by adding 750 µl of acetic acid. Finally, 250 µl of ninhidryn will be added to the samples followed by incubation at 95°C for one hour. The activity of the arginase present per sample will be detected by the conversion of L-arginine to L-ornithine by colorimetric assay at 570 nm using a standard curve of known concentrations of L-ornithine.
  Arginase I levels. Arginase I levels will be tested in plasma of study volunteer donors using an ELISA kit (BioVendor), following the vendor's protocols.
myeloid-derived suppressor cells (MDSC) | Baseline clinical visit
  MDSC will be isolated and characterized as described before, by using CD14-negative selection and CD11b-positive selection magnetic beads (Miltenyi Biotech) or by labeling PBMC with anti-CD66b followed by anti-FITC magnetic bead separation, according to the manufacturer's specifications. Additional markers will include CD33, and CD15. Morphology of the cells (MDSC and PMN) will be performed by staining of cytospins. Briefly, 5 × 104 cells will be centrifuged in a StatSpin CytoFuge centrifuge at 8.5 × g for 4 min and stained using Harleco Hemacolor kit from EMD. . Flow cytometry will also be used to determine the percentage of monocytic or granulocytic MDSC using several fluorescence-labeled antibodies, including anti-CD11b, CD14, CD15, CD33, CD66 and HLA-DR.
Serum inflammatory markers change | Baseline visit and and post intervention at 13 to 15 weeks
  Serum inflammatory markers will be obtained by simple blood draw and evaluated by Enzyme Linked Immunoassay (ELISA); the panel will measure 11 pro- and anti-inflammatory factors and cytokines previously shown to be associated with inflammatory diseases (gastritis or prostate cancer), with asthma, or with obesity. These include: Adiponectin, IL13~IL5, Leptin, TGFp, Arginase 1, IL-6, ILIO, PGE2, C-Reactive Protein, IL3, TNFa, IL4.
HbA1C (Hemoglobin A1C or Glycosylated hemoglobin change | Baseline visit and and post intervention at 13 to 15 weeks
  HbA1C will be measured in plasma and blood to evaluate blood sugar levels.
Lipid profile change | Baseline visit and and post intervention at 13 to 15 weeks
  total cholesterol, high density lipoprotein, low density lipoprotein, triglycerides will be measured in plasma
HOMA-IR (homeostasis model assessment-estimated insulin resistance change | Baseline visit and and post intervention at 13 to 15 weeks
  HOMA-IR is a measure to determine the degree of insulin resistance as a marker for general homeostasis. To determine this index, levels of fasting insulin and glucose will be obtained from blood samples drawn for the lipid profile analysis described above, which will determine whether cholesterol and two of the other chemicals in the blood sample, e.g. insulin and glucose, are related to the inflammation seen in obese asthmatic children. To calculate the HOMA-IR we will use the following formula: fasting glucose (mmol/L) x fasting insulin (mIU/L)/22.5.
Weight in kilograms | Baseline visit and and post intervention at 13 to 15 weeks
  Weight in kilograms will be obtained by standardized scale and weight values will be evaluated using standard National Center for Health Statistics (NCHS) growth charts.
Height in centimeters | Baseline visit and and post intervention at 13 to 15 weeks
  Height will be measured using stadiometer and evaluated by standard National Center for Health Statistics (NCHS) growth charts.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda S Sothern, PhD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No